CLINICAL TRIAL: NCT04893083
Title: A Multi-center, Non-interventional Phase 0 Study for the Collection of Biospecimens From Patients With Parkinson's Disease.
Brief Title: A Non-interventional Study for the Collection of Biospecimens From Patients With Parkinson's Disease
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Neuron23 Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: N23-PD-001
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LRRK2 Mutant PD: Patients with a G2019S mutation
- LRRK2 Wild Type PD Low burden: Patients with a low burden of genetic modifiers
- LRRK2 Wild Type High burden: Patients with a high burden of genetic modifiers

SUMMARY:
This study aims to collect, analyze and preserve biospecimens from patients with or without LRRK2-associated Parkinson's Disease for the purpose of discovering and developing new treatments and novel biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥40
* Clinical diagnosis of Parkinson's disease meeting United Kingdom Brain Bank criteria and modified Hoehn and Yahr Stage I, II, or III;
* Willing to undergo genetic testing for neurologic genotyping panel; -If being treated for Parkinson's disease, must have been on a stable dose of anti- Parkinson's disease medications for a minimum of 30 days prior to Day 1;
* If taking statins, fibrates, antipsychotic or anticonvulsant medications at Day 1, must have been on a stable dose for a minimum of 30 days, and are not likely to require a change in dosage for the remainder of the study;

Exclusion Criteria:

* Any major medical illness or unstable medical condition within 6 months of screening that, in the opinion of the Investigator or Sponsor, may interfere with the subject's ability to comply with study procedures or abide by study restrictions.
* Diagnosis of a significant central nervous system disease other than Parkinson's disease(eg, Huntington's disease, frontotemporal dementia, multi-infarct dementia, normal pressure hydrocephalus, multiple system atrophy, progressive supranuclear palsy, drug- induced parkinsonism, Alzheimer's disease)
* History of stroke;
* History of epilepsy or seizure disorder other than febrile seizures as a child, or any seizure or unexpected loss of consciousness (eg, syncope) within 6 months prior to Day 1;
* History of traumatic brain injury with residual neurological deficit; -If taking anti-Parkinson's disease medication(s)and are likely to require a change in anti- Parkinson's disease medication(s) during the study;
* Known active infectious disease or active infections within 30 days prior to Day 1;
* Any vaccination within 21 days prior to Day 1;
* Currently taking, or planning to take, anti-coagulant medications or antiplatelet medications during the study;
* Allergy to Lidocaine (xylocaine) or its derivatives or any other LP contraindications;
* Any other condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the Investigator, unacceptably increase the subject's risk by participating in the study; -Any systemic glucocorticoids taken within 14 days prior to Day 1 or non-steroidal anti- inflammatory drugs taken within 4 days prior to Day 1;
* Received blood products within 30 days prior to Day 1;
* Donated blood within 30 days prior to Day 1.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients will be recruited across this multi-center, global clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Genetic Marker | 1 day
  Test for LRRK2 mutations in Parkinson disease patients; identifying patients with potential genetic modifiers

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Quest Research Institute, Farmington Hills, Michigan
  - Evergreen Health, Kirkland, Washington
- Canada (2):
  - Universite Laval, Québec, Quebec
  - McGill University, Montreal
- Assistance Publique - Hospitaux de Paris, Paris, France
- Israel (2):
  - Sheba Tel HaShomer, Ramat Gan
  - Tel Aviv Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No